CLINICAL TRIAL: NCT04106258
Title: A Pilot Study of Hemoporfin Photodynamic Therapy in Children (2-7 Years Old) With Port-wine Stain
Brief Title: A Pilot Study of Hemoporfin PDT in Children(2-7 Years Old) With Port-wine Stain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: HMME-C1904
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Port-wine Stain
MeSH Terms: conditions — Port-Wine Stain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low light dose (Experimental): PDT is applied to the patients at low light dose : power density of 60mW/cm2 for 20 minutes
  Interventions: Drug: Hemoporfin PDT
- high light dose (Experimental): PDT is applied to the patients at high light dose : power density of 75mW/cm2 for 20 minutes
  Interventions: Drug: Hemoporfin PDT

INTERVENTIONS:
Drug: Hemoporfin PDT — Photodynamic therapy is performed using hemoporfin under general anesthesia. Hemoporfin（5mg/kg）is infused for 20 minutes, followed by light illumination at 10 minutes from the start of infusion. Different light dose of PDT is applied to the patients.

SUMMARY:
This pilot study aims to evaluate the safety and efficacy of hemoporfin photodynamic therapy (PDT) with different light doses for port-wine stain (PWS）in 2-7 years old children. The pharmacokinetic behavior and pharmacokinetic parameters of hemoporfin in children will be investigated as well.

ELIGIBILITY:
Inclusion Criteria:

* Children with clinical diagnosis of PWS；
* ≥2 years old and <7 years old；
* The guardians agreed to voluntarily participate in this study and signed the informed consent agreement

Exclusion Criteria:

* Therapy area located outside of head and neck;
* Other skin diseases that might interfere with the efficacy evaluation;
* Patients with respiratory disease, severe pulmonary dysfunction, history of airway hyperresponsiveness, or family history of suspected malignant hyperthermia;
* Preexist scars in the treatment area caused by previous treatment, which might interfere with the efficacy and safety evaluation;
* with allergic diseases; known to be allergic to eggs, milk or soy protein; known to have skin photoallergies, porphyria or known allergic history of experimental drugs (porphyrins) and chemically structure similar drugs; known allergic history of anesthetics; allergic constitution;
* Cicatricial constitution;
* Immunocompromised conditions or need long-term use of glucocorticoids and immunosuppressive agents;
* Electrocardiographic abnormalities or organic heart diseases;
* Hepatic or renal functions abnormal (alanine aminotransferase or aspartate transaminase or total bilirubin > 1.5 upper limit of normal [ULN], or serum creatinine or blood urea nitrogen > 1.5 ULN);
* Coagulation disorders;
* Patients with severe neurological, psychiatric, endocrine and cardiovascular diseases; with epilepsy history or recent epileptic seizures;
* Be evaluated not suitable for anaesthesia by risk assessment before anaesthesia；
* Previous therapy of PWS within the last 4 weeks;
* Participation in any clinical studies within the last 4 weeks;
* Be judged not suitable to participate the study by the investigators

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Response rate | week 8
  proportion of patients achieving at least some improvement (color blanching from the baseline >= 20%)
Incidence of adverse events and adverse reactions | up to 24 weeks after the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No